CLINICAL TRIAL: NCT05936099
Title: Development and Implementation of a Tobacco and ENDS Use Intervention for Adolescents and Young Adults in the Pediatric Hospital
Brief Title: Adolescent Inpatient Tobacco and ENDS Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Abbey Masonbrink, Pediatric Hospitalist, MD MPH, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002116; K23DA055736 (NIH)
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Vaping; Smoking
Keywords: Vaping; Adolescents; Cessation
MeSH Terms: conditions — Vaping; Smoking | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will complete the baseline survey and receive an informational brochure
- Intervention (Experimental): Participants will complete the baseline survey, receive a behavioral health intervention supported by computerized decision support, and take an exit survey
  Interventions: Behavioral: E-cigarette & Tobacco Use Treatment Intervention

INTERVENTIONS:
Behavioral: E-cigarette & Tobacco Use Treatment Intervention — The behavioral intervention includes health education on vaping health risk and outcomes, motivational interviewing, and assisted quit planning from a health educator and counseling and nicotine replacement therapy (if appropriate) provided by a physician.
  Arms: Intervention

SUMMARY:
The purpose of this study is to develop and evaluate an evidence-based intervention to assist adolescents and young adults with current vaping to quit vaping and smoking.

DETAILED DESCRIPTION:
Use of electronic nicotine delivery system (ENDS), which are noncombustible tobacco products (e.g., e-cigarettes), has increased dramatically among youth and is associated with numerous adverse health outcomes as well as use of alcohol and other illicit substances. National guidelines recommend counseling to address tobacco use at every adolescent clinical visit; however, many at-risk adolescents do not routinely attend primary care. Although evidence supports treatment of tobacco use during an adult hospitalization, no interventions have been developed or tested in the pediatric hospital setting. Based on promising theoretically-based evidence from the primary care and hospital settings, we will design, iteratively refine and assess implementation of a novel tobacco and ENDS use intervention for hospitalized adolescents and young adults (AYAs). We do so by conducting a randomized controlled pilot study (n=144) with 3-month follow up to evaluate preliminary efficacy as well as implementation outcomes (i.e., acceptability, feasibility, fidelity).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital
* Screens positive for past 30 day e-cigarette use
* Parent/guardian agrees to leave the room

Exclusion Criteria:

* Age is less than 14 years or over 21 years
* Not comfortable speaking/reading English
* Too ill to participate
* Severe psychiatric illness
* Too developmentally delayed/cognitively impaired

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbey Masonbrink, MD, MPH, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wooten S, Catley D, Miller MK, Wilson K, Richter KP, Masonbrink A. Treatment of e-cigarette use among hospitalised adolescents and young adults: a protocol for intervention development and evaluation of preliminary efficacy and implementation outcomes in a randomised controlled trial. BMJ Open. 2025 Jan 8;15(1):e094323. doi: 10.1136/bmjopen-2024-094323. PMID 39779271

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 48 | 96
Completed | 38 | 58
Not Completed | 10 | 38
Not completed — Lost to Follow-up | 10 | 38

BASELINE CHARACTERISTICS:
Population: All enrolled participants completed the baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 48 | 96 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (1.3) | 16.2 (1.3) | 16.2 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 63 | 94
  Male | 17 | 33 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 15 | 25
  Not Hispanic or Latino | 35 | 80 | 115
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 17 | 24
  White | 27 | 56 | 83
  More than one race | 9 | 16 | 25
  Unknown or Not Reported | 5 | 4 | 9
Past 30 day e-cigarette use [Count of Participants; unit: Participants] — Potential participants were pre-screened for recent (past 30 day) use of e-cigarettes
  Participants
    0 Days | 0 | 0 | 0
    1-5 days (occasional) | 18 | 31 | 49
    6-19 days (intermittent) | 12 | 24 | 36
    20+ days (frequent) | 16 | 40 | 56
    Missing | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Self-reported 30-day Abstinence
Description: Self reported cessation, assessed at 3 month follow up survey.
Time Frame: 3 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 38 | 58
Participants | 16 | 25
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.91, Fisher Exact
Statistical Analysis 2: Comparison: Intervention; Intent-to-treat sensitivity analysis to assess the odds of tobacco abstinence in the intervention arm when compared to the control arm; Test type: Other; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.27 to 2.19]

2. Primary Outcome: Biochemically Verification of Past 30 Day Cessation
Description: For participants who self-reported past 30 day cessation, an option was provided to biochemically verify cessation with a mailed saliva sample.
Time Frame: 3 month follow-up
Population: Only those who indicated they had not used tobacco in any form (traditional cigarettes or electronic cigarettes) and had not taken nicotine replacement therapy (NRT) in the past 30 days were given the option to complete the biochemical verification.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 58 | 38
Participants
  Agreed to do biochemical verification & successfully completed test | 1 | 2
  Agreed to do biochemical verification & did not complete test | 5 | 2
  Declined offer to complete biochemical verification test | 16 | 10
  Ineligible for to complete biochemical verification test due to tobacco use or NRT use | 36 | 24

3. Secondary Outcome: Acceptability of Intervention - Satisfaction and Likeliness to Recommend Program
Description: Ratings from participants on perceived acceptability (i.e., satisfaction and usefulness) of the intervention
Time Frame: Study completion (approximately 12 weeks)
Population: This outcome measure was assessed following the index intervention session so all 96 enrolled intervention participants completed this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 96
Participants
  Satisfaction with the intervention: Not at all satisfied / Extremely unlikely | 0
  Satisfaction with the intervention: A little satisfied / Unlikely | 3
  Satisfaction with the intervention: Not sure satisfied / Neutral | 8
  Satisfaction with the intervention: Somewhat satisfied / Likely | 34
  Satisfaction with the intervention: Very satisfied / Extremely likely | 51
  Likely to recommend the intervention to friends or family: Not at all satisfied / Extremely unlikely | 1
  Likely to recommend the intervention to friends or family: A little satisfied / Unlikely | 3
  Likely to recommend the intervention to friends or family: Not sure satisfied / Neutral | 20
  Likely to recommend the intervention to friends or family: Somewhat satisfied / Likely | 37
  Likely to recommend the intervention to friends or family: Very satisfied / Extremely likely | 35

4. Secondary Outcome: Acceptability of Intervention - Utility of Intervention
Description: Acceptability of the intervention assessed by intervention element completion rates (i.e. overall uptake of support resources).
Time Frame: Study completion (approximately 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 96
Participants
  Made a quit plan during the index session | 47
  Were interested in nicotine replacement therapy during the index session | 14
  Were prescribed nicotine replacement therapy during the index session | 11
  Enrolled in a text-to-quit program during the index session | 13
  Were provided addiction resources information during the index session | 67

5. Secondary Outcome: Feasibility of Intervention - Duration of Intervention
Description: Assessment of the feasibility of the intervention based on information about delivery gathered from the computerized decision making system (CDS) such as the duration of the intervention.
Time Frame: Study completion (approximately 12 weeks)
Population: This outcome measure was assessed for the intervention arm only.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intervention
Number analyzed (Participants) | 96
minutes | 32 [28 to 39]

6. Secondary Outcome: Feasibility of Intervention - Intervention Interruptions
Description: Assessment of the feasibility of the intervention based on information about delivery gathered from the computerized decision making system (CDS) such as the number of interruptions (by clinical staff, parents, or others) that occurred during intervention delivery.
Time Frame: Study completion (approximately 12 weeks)
Population: This outcome measure was assessed for the intervention arm only.
Measure: Median (Inter-Quartile Range); unit: number of interruptions
Arm/Group | Intervention
Number analyzed (Participants) | 96
number of interruptions | 0 [0 to 5]

7. Secondary Outcome: Feasibility of Intervention - Health Educator Survey
Description: Feasibility of the intervention as assessed by the health educator who delivered the intervention.
Time Frame: Study completion (approximately 12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 96
Participants
  Agreed/ Strongly Agreed the intervention was easy to deliver | 95
  Agreed/Strongly Agreed there was enough time to deliver the intervention | 94

8. Secondary Outcome: Fidelity of Intervention Delivered by a Health Educator
Description: Extent of fidelity achieved in intervention delivery by a health educator. The mean score was calculated from 0 (never/very poor) to 5 (always/very good) for each of the 10 fidelity rating questions, which were summed, with a maximum possible score of 50. The scale utilized was an adapted version of the Motivational Interviewing Treatment Integrity tool (MITI).
Time Frame: Study completion (approximately 12 weeks)
Population: Recordings of intervention sessions were randomly selected at set intervals during the enrollment period and scored.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 13
scores on a scale | 43 (3.1)

ADVERSE EVENTS:
Time Frame: From enrollment to the end of 3 month follow up
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/96
Other Adverse Events (participants affected / at risk) | 0/48 | 0/96

LIMITATIONS AND CAVEATS:
We enrolled e-cigarette users at any stage of motivation to quit, which may have impacted intervention efficacy. Due to practical limitations participants and the research team were not blinded to study conditions which may have led to bias in the assessment of outcome. We relied on self-report which is susceptible to social desirability bias and had very low biochemical verification completion rates to confirm our primary outcome. As a single site study there is limited generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT05936099/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT05936099/SAP_001.pdf